CLINICAL TRIAL: NCT00813709
Title: Double-blind Extension of the Study 27025 (REFLEX) to Obtain Long-term Follow-up Data in Patients With Clinically Definite MS and Patients With a First Demyelinating Event at High Risk of Converting to MS, Treated With Rebif® New Formulation (REFLEXION)
Brief Title: Long-term Follow-Up of Patients Who Participated in Study 27025 (REFLEX)
Acronym: REFLEXION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28981
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Interferon 1-beta; Clinical Definite Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- RNF 44 mcg thrice weekly (Active Comparator)
  Interventions: Drug: RNF
- RNF 44 mcg once weekly and placebo (Active Comparator)
  Interventions: Drug: RNF; Drug: Placebo
- Placebo/RNF 44 mcg thrice weekly (Active Comparator)
  Interventions: Drug: RNF

INTERVENTIONS:
Drug: RNF — Single dose of RNF will be administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months.
  Other Names: Rebif®
  Arms: RNF 44 mcg thrice weekly
Drug: RNF — Single dose of RNF will be administered subcutaneously once weekly at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months.
  Other Names: Rebif®
  Arms: RNF 44 mcg once weekly and placebo
Drug: RNF — Participants who were initially randomized in Study 27025 (REFLEX) to the placebo treatment group will be switched to single dose of RNF administered subcutaneously three times weekly at least 48 hours apart at a dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months.
  Other Names: Rebif®
  Arms: Placebo/RNF 44 mcg thrice weekly
Drug: Placebo — Single dose matching placebo will be administered subcutaneously twice weekly. Placebo is supplied as a transparent, sterile solution for injection in pre-filled syringes matching the RNF pre-filled syringes, each containing 0.5 milliliter (mL).
  Arms: RNF 44 mcg once weekly and placebo

SUMMARY:
REFLEXION is a double blind extension of the study 27025 (NCT00404352) (REFLEX). The purpose of the study is to obtain long-term follow-up data in subjects with clinically definite multiple sclerosis (MS) and subjects with a first demyelinating event at high risk of converting to MS, treated with fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of interferon [IFN]-beta-1a (RNF).

DETAILED DESCRIPTION:
The objective of the study is to investigate whether RNF treatment initiated after the first clinical event versus delayed treatment results in the prolongation of time to Clinically Definite Multiple Sclerosis (CDMS) conversion up to Month 36 and up to Month 60 since randomization in Study 27025 (REFLEX). Furthermore, the study is intended to explore whether RNF treatment initiated after the first clinical event versus delayed treatment delays disability (including development of secondary progressive MS) and reduces disease activity (including the annual relapse rate [ARR]) in the long term (up to Month 36 and up to Month 60 since randomization in Study 27025 (REFLEX). The study will also assess the long-term safety profile of RNF (up to Month 36 and up to Month 60 since randomization in Study 27025 (REFLEX).

ELIGIBILITY:
Inclusion Criteria:

* Reach scheduled end of study in Study 27025 (REFLEX) (completion of 24 months participation)
* Medical assessment by the Investigator/treating physician from study 27025 that there is no objection to the subject's participation in this extension trial considering the medical experience from Study 27025 (REFLEX). Special attention should be given to laboratory abnormalities and clinically significant liver, renal and bone-marrow dysfunction
* If female, subject must:

  * be neither pregnant nor breast-feeding, nor attempting to conceive
  * use a highly effective method of contraception. A highly effective method of contraception is defined as those which result in a low failure rate (that is [i.e.] less than 1 percent [%] per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner
* Subject is willing to follow study procedures
* Subject has given written informed consent

Exclusion Criteria:

* Subject has any disease other than MS that could better explain the subject's signs and symptoms
* Subject has a primary progressive course of MS
* Subject has total bilirubin greater than 2.5 times upper limit of normal (ULN) at both Month 24 and at the previous visit (i.e. Month 21) (subjects with greater than 2.5 times ULN at Month 24 only are eligible for enrollment and should be managed as per label recommendations until normalization of the value)
* Subject has total aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or alkaline phosphatase (ALP) greater than 2.5 times the ULN values at both Month 24 and at the previous visit (i.e. Month 21) (subjects with greater than 2.5 times ULN at Month 24 only are eligible for enrollment and should be managed as per label recommendations until normalization of the value)
* Subject suffers from another current autoimmune disease
* Subject suffers from major medical or psychiatric illness (including history of, or current, severe depressive disorders and/or suicidal ideation) that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
* Subject has a history of seizures not adequately controlled by treatment
* Subject has cardiac disease, such as angina, congestive heart failure or arrhythmia
* Subject has a known allergy to IFN-beta or the excipient(s) of the study medication
* Subject has any condition that could interfere with the MRI evaluation
* Subject has a known allergy to gadolinium-diethylene triamine pentaacetic acid (DTPA)
* Subject has a history of alcohol or drug abuse
* Subject has previously participated in this study
* Subject has moderate to severe renal impairment
* Subject is pregnant or lactating
* Subject has any medical, psychiatric or other conditions that compromise his/her ability to understand the subject information, to give informed consent, to comply with the study protocol, or to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.A., Geneva
Locations (57):
- Research Site, Mendoza, Argentina
- Research Site, Graz, Austria
- Belgium (2):
  - Research Site, Bruges
  - Research Site, Leuven
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
- Canada (2):
  - Research Site, Ontario
  - Research Site, Victoria British Columbia
- Croatia (5):
  - Research Site, Karlovac
  - Research Site, Osijek
  - Research Site, Rijeka
  - Research Site, Split
  - Research Site, Zagreb
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Research Site, Oulu, Finland
- France (2):
  - Research Site, Paris
  - Research Site, Poissy
- Germany (2):
  - Research Site, Hanover
  - Research Site, Henningsforf
- Research Site, Athens, Greece
- Israel (2):
  - Research Site, Safed
  - Research Site, Tel Litwinsky
- Italy (2):
  - Research Site, Milan
  - Research Site, Padua
- Research Site, Riga, Latvia
- Research Site, Beirut, Lebanon
- Research Site, Rabat, Morocco
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Lisbon, Portugal
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (7):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Veliky Novgorod
  - Research Site, Yekaterinburg
- Serbia (2):
  - Reserch Site, Belgrade
  - Research Site, Niš
- Research Site, Prešov, Slovakia
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Madrid
  - Research Site, Seville

REFERENCES:
- [Derived] Comi G, De Stefano N, Freedman MS, Barkhof F, Uitdehaag BM, de Vos M, Marhardt K, Chen L, Issard D, Kappos L. Subcutaneous interferon beta-1a in the treatment of clinically isolated syndromes: 3-year and 5-year results of the phase III dosing frequency-blind multicentre REFLEXION study. J Neurol Neurosurg Psychiatry. 2017 Apr;88(4):285-294. doi: 10.1136/jnnp-2016-314843. Epub 2016 Dec 30. PMID 28039317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were randomized in Study 27025 (NCT00404352) were eligible to enroll into extension Study 28981 (NCT00813709) whether or not they completed main study on Investigational Medicinal Product (IMP), or no treatment or received other disease-modifying drugs (DMDs) during course of main study. No re-randomization was done for this study.
Pre-assignment Details: 517 participants randomized in Study 27025 used in this study as integrated intention to treat (ITT) population. Out of the 517, 402 participants took part in study 28981: 300 comprised the double blind (DB) population and 122 comprised the open label (OL) population (some participants (20) were included in both populations)
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (DB Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN]-beta-1a (RNF) injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first.
- RNF 44 Mcg Once Weekly (DB Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first.
- RNF 44 Mcg Thrice Weekly (DB Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first.
- Placebo/RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly: Participants after having converted to CDMS during study 28981 (REFLEXION), received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. The participants who were converted to CDMS in study 27025 (REFLEX) and were enrolled in this study continued receiving RNF 44 mcg three times weekly until 60 months.
- RNF 44 Mcg Once Weekly /OL RNF 44 Mcg Thrice Weekly; RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly: Participants after having converted to CDMS during study 28981 (REFLEXION), received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. The participants who were converted to CDMS in study 27025 (REFLEX) and were enrolled in this study continued receiving RNF 44 mcg three times weekly until 60 months.
Period: Double Blind Period
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) | RNF 44 Mcg Once Weekly (DB Population) | RNF 44 Mcg Thrice Weekly (DB Population) | Placebo/RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly | RNF 44 Mcg Once Weekly /OL RNF 44 Mcg Thrice Weekly | RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly
Started | 84 | 117 | 99 | 0 | 0 | 0
Treated | 83 | 114 | 98 | 0 | 0 | 0
Completed | 53 | 76 | 68 | 0 | 0 | 0
Not Completed | 31 | 41 | 31 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 2 | 0 | 0 | 0
Not completed — Switched to open label phase | 9 | 26 | 18 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 3 | 1 | 0 | 0 | 0
Not completed — Other | 14 | 9 | 6 | 0 | 0 | 0
Period: Open Label Period
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) | RNF 44 Mcg Once Weekly (DB Population) | RNF 44 Mcg Thrice Weekly (DB Population) | Placebo/RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly | RNF 44 Mcg Once Weekly /OL RNF 44 Mcg Thrice Weekly | RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly
Started | 0 | 0 | 0 | 58 (49 participants in OL period initially + 9 participants from DB converted to CDMS during the study) | 51 (25 participants in OL period initially + 26 participants from DB converted to CDMS during the study) | 46 (28 participants in OL period initially + 18 participants from DB converted to CDMS during the study)
Treated | 0 | 0 | 0 | 57 | 51 | 45
Completed | 0 | 0 | 0 | 38 | 41 | 35
Not Completed | 0 | 0 | 0 | 20 | 10 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 4 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3 | 1 | 1
Not completed — Randomized but not treated | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 11 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Baseline data was presented for ITT population (402 participants) which included participants who had completed the REFLEX Study 27025 (NCT00404352) and were enrolled in this extension Study 28981 (REFLEXION).
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (ITT Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of RNF injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months. 84 participants were initially assigned to DB RNF 44 mcg thrice weekly and 49 participants were initially assigned to OL RNF 44 mcg thrice weekly (9 participants from DB converted to CDMS and switched to OL period over course of this study)
- RNF 44 Mcg Once Weekly (ITT Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. 117 participants were initially assigned to DB RNF 44 mcg thrice weekly and 25 participants were initially assigned to OL RNF 44 mcg thrice weekly (26 participants from DB converted to CDMS and switched to OL period over course of this study)
- RNF 44 Mcg Thrice Weekly (ITT Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. 99 participants were initially assigned to DB RNF 44 mcg thrice weekly and 28 participants were initially assigned to OL RNF 44 mcg thrice weekly (18 participants from DB converted to CDMS and switched to OL period over course of this study)
- Total: Total of all reporting groups
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (ITT Population) | RNF 44 Mcg Once Weekly (ITT Population) | RNF 44 Mcg Thrice Weekly (ITT Population) | Total
Number analyzed (Participants) | 133 | 142 | 127 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (8.2) | 31.4 (8.2) | 31.8 (8.6) | 31.4 (8.3)
Age, Customized [Number; unit: participants]
  Less than 30 years | 67 | 66 | 55 | 188
  Greater than or equal to 30 years | 66 | 76 | 72 | 214
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 88 | 78 | 248
  Male | 51 | 54 | 49 | 154
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 0 | 1 | 0 | 1
  White | 133 | 141 | 127 | 401

OUTCOME MEASURES:

1. Primary Outcome: Time to Conversion to Clinically Definite Multiple Sclerosis (CDMS) Defined by Either a Second Attack or a Sustained Increase (Greater Than or Equal to 1.5 Points) in the Expanded Disability Status Scale (EDSS) Score up to 36 Months
Description: CDMS was defined by the occurrence of a second attack or relapse over 36 months in participants who presented with clinically isolated syndrome (CIS) accompanied by an abnormal magnetic resonance imaging (MRI) scan. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]) was calculated. Time to conversion to CDMS was represented by Kaplan-Meier estimates of the cumulative percentage (%) of participants with CDMS.
Time Frame: Baseline (Day 1 of Study 27025) up to 36 Months
Population: Data has been presented as per planned analysis for integrated ITT population which included all participants who were randomized in REFLEX study 27025 (NCT00404352).
Measure: Number (95% Confidence Interval); unit: Cumulative % of participants with CDMS
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN]-beta-1a (RNF) injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first. After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months.
- RNF 44 Mcg Once Weekly (Integrated ITT Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months.
- RNF 44 Mcg Thrice Weekly (Integrated ITT Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months.
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
Cumulative % of participants with CDMS | 41.3 [33.5 to 49.1] | 27.6 [20.6 to 34.6] | 27.1 [19.9 to 34.3]
Statistical Analysis 1: Comparison: Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) vs RNF 44 Mcg Thrice Weekly (Integrated ITT Population); Test type: Superiority or Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 0.555, 95% CI 2-sided [0.378 to 0.816]
Statistical Analysis 2: Comparison: Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) vs RNF 44 Mcg Once Weekly (Integrated ITT Population); Test type: Superiority or Other; p = 0.006, Log Rank; Hazard Ratio (HR) = 0.573, 95% CI 2-sided [0.391 to 0.839]
Statistical Analysis 3: Comparison: RNF 44 Mcg Once Weekly (Integrated ITT Population) vs RNF 44 Mcg Thrice Weekly (Integrated ITT Population); Test type: Superiority or Other; p = 0.941, Log Rank; Hazard Ratio (HR) = 0.993, 95% CI 2-sided [0.654 to 1.510]

2. Secondary Outcome: Time to Confirmed Expanded Disability Status Scale (EDSS) Progression up to 36 Months
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. A confirmed EDSS progression was defined EDSS greater than or equal to 1.0 point confirmed during a visit performed 6 months later. Time to confirmed EDSS progression was represented by Kaplan-Meier estimates of the cumulative percentage (%) of participants with confirmed EDSS progression.
Time Frame: Baseline (Day 1 of Study 27025) up to 36 Months
Population: as for outcome 1
Measure: Number; unit: % of participants with EDSS progression
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
% of participants with EDSS progression | 7.5 | 11.8 | 13.2
Statistical Analysis 1: Comparison: Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) vs RNF 44 Mcg Thrice Weekly (Integrated ITT Population); Test type: Superiority or Other; p = 0.205, Log Rank
Statistical Analysis 2: Comparison: Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) vs RNF 44 Mcg Once Weekly (Integrated ITT Population); Test type: Superiority or Other; p = 0.263, Log Rank
Statistical Analysis 3: Comparison: RNF 44 Mcg Once Weekly (Integrated ITT Population) vs RNF 44 Mcg Thrice Weekly (Integrated ITT Population); Test type: Superiority or Other; p = 0.629, Log Rank

3. Secondary Outcome: Number of Combined Unique Active (CUA) Lesions, New Time Constant 2 (T2) Lesions, New Gadolinium Enhanced (Gd+) Lesions and New Time Constant 1 (T1) Lesions Per Participant Per Scan at Month 36
Description: Number of CUA lesions, new T2 lesions, new Gd+ lesions and new T1 lesions were measured by using MRI scans.
Time Frame: Month 36
Population: Data has been presented as per planned analysis for integrated ITT population which included all participants who were randomized in REFLEX study 27025 (NCT00404352). 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure at this time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 124 | 133 | 114
lesions
  CUA Lesions | 1.02 (1.85) | 1.83 (3.317) | 1.63 (5.947)
  New T2 Lesions | 0.83 (1.545) | 1.39 (2.573) | 1.19 (4.217)
  New Gd+ Lesions | 0.17 (0.506) | 0.40 (1.354) | 0.41 (1.754)
  New T1 Lesions | 0.69 (1.721) | 1.09 (2.482) | 0.91 (4.143)

4. Secondary Outcome: Change From Baseline in Time Constant 1 (T1) Hypointense Lesion Volume and Time Constant 2 (T2) Lesion Volume at Month 36
Description: Change from baseline in lesion volume was measured by using MRI scans for T1 hypointense lesions and T2 lesions at Month 36
Time Frame: Baseline (Day 1 of Study 27025), Month 36
Population: Data has been presented as per planned analysis for integrated ITT population which included all participants who were randomized in REFLEX study 27025 (NCT00404352). "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
cubic millimeter (mm^3)
  T1 lesion volume at Baseline (n=171,175,171) | 670.3 (1054.1) | 774.8 (1288.0) | 675.0 (1049.9)
  T1 lesion volume Change: Month 36(n=124,133,114) | 303.2 (1034.6) | 272.0 (921.4) | 133.3 (763.5)
  T2 lesion volume at Baseline (n=171,175,171) | 3334.9 (3990.4) | 3853.1 (4716.7) | 3110.5 (3410.7)
  T2 lesion volume Change: Month 36(n=124,133,114) | -3.8 (2101.8) | -56.9 (2436.3) | -398.1 (1415.4)

5. Secondary Outcome: Percent Change From Baseline in Brain Volume at Month 36
Description: Percent change in brain volume was measured by using MRI scans.
Time Frame: Baseline (Day 1 of Study 27025), Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 120 | 132 | 112
percent change | -1.02 (1.248) | -0.86 (1.073) | -1.14 (1.321)

6. Secondary Outcome: Percentage of Participants With Conversion to McDonald Multiple Sclerosis (MS) up to 36 Months
Description: The McDonald criteria use dissemination in time and space established by MRI findings to provide a clinical diagnosis for MS. Dissemination in time is established by a new T2 or Gd+ lesion found on a repeat MRI. Dissemination in space is established by the presence of any 3 of the following: 1 Gd+ lesion or 9 T2 bright lesions if there is no enhancement; greater than or equal to 1 infratentorial lesion; greater than or equal to 1 juxtacortical lesion; greater than or equal to 3 periventricular lesions.
Time Frame: Baseline (Day 1 of Study 27025) up to CDMS conversion and/or up to 36 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
percentage of participants | 84.2 | 76.0 | 66.7

7. Secondary Outcome: Change From Baseline in Paced Auditory Serial Addition Test 3 (PASAT-3) Score at Month 36
Description: The Paced Auditory Serial Addition Test (PASAT) is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Score ranges from '0-60'. Higher scores reflect better neurological function and a positive change from baseline indicates improvement.
Time Frame: Baseline (Day of Study 27025), Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
units on a scale
  Baseline (n=171,175,171) | 0.0358 (0.8787) | -0.0909 (1.1223) | 0.0031 (1.1387)
  Change at Month 36 (n=123,135,118) | 0.3483 (0.6949) | 0.5044 (0.7588) | 0.4515 (0.9164)

8. Secondary Outcome: Percentage of Relapse-Free Participants at Month 36
Description: A relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, lasting for 24 hours and with a previous period for more than 30 days with a stable or an improving condition.
Time Frame: Month 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
Percentage of participants | 42.7 | 58.3 | 51.5

9. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Month 36
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. The change in EDSS score at Month 36 was calculated as EDSS score at Month 36 minus EDSS score at baseline.
Time Frame: Baseline (Day of Study 27025), Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
units on a scale
  Baseline (n=171,175,171) | 1.53 (0.77) | 1.50 (0.72) | 1.51 (0.83)
  Change at Month 36 (n=120,136,116) | -0.21 (0.93) | -0.11 (0.96) | -0.09 (0.90)

10. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score at Month 36
Description: The MSFC is a multidimensional clinical outcome measure which consists of three sub-tests; Timed 25-Foot Walk, 9-Hole Peg Test and Paced Auditory Serial Addition Test-3(PASAT-3). The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The 9-Hole Peg Test is a quantitative measure of upper extremity (arm and hand) function. The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Standardized results (Z-scores) of these sub-tests and the overall MSFC Z-score as an average of these three Z-scores was calculated. Higher Z-scores reflect better neurological function and a positive change from baseline indicates improvement. An increase in score indicates an improvement (range -3 to +3).
Time Frame: Baseline (Day 1 of Study 27025), Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
Z-score
  MFSC score at Baseline (n=171,175,171) | 0.0352 (0.5844) | 0.0071 (0.6653) | -0.0575 (0.6226)
  Change at Month 36 (n=123,135,118) | 0.1993 (0.4863) | 0.2529 (0.5794) | 0.3074 (0.6071)

11. Secondary Outcome: Numbers of Participants With Binding Antibodies (BAb) and Neutralizing Antibody (NAb) at Month 36
Description: BAbs are all antibodies which are capable of binding to the investigational drug molecule (RNF) irrespective of their binding site. NAbs are defined as a subgroup of BAbs which bind to the active sites of the RNF and therefore neutralize its potency. NAbs were detected using a viral cytopathic assay. BAbs were measured by using an ELISA (Enzyme-linked immunosorbent assay).
Time Frame: Month 36
Population: Data has been presented as per planned analysis for integrated DB population which included all participants who received at least one dose of DB treatment in REFLEX study 27025 (NCT00404352). 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure at this time point.
Measure: Number; unit: participants
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (Integrated DB Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN]-beta-1a (RNF) injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first.
- RNF 44 Mcg Once Weekly (Integrated DB Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first.
- RNF 44 Mcg Thrice Weekly (Integrated DB Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first.
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated DB Population) | RNF 44 Mcg Once Weekly (Integrated DB Population) | RNF 44 Mcg Thrice Weekly (Integrated DB Population)
Number analyzed (Participants) | 118 | 131 | 118
participants
  BAb- | 77 | 97 | 88
  BAb+ | 41 | 34 | 30
  NAb- | 100 | 109 | 99
  NAb+ | 18 | 22 | 19

12. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Treatment Discontinuation
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. SAE: Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition.
Time Frame: Month 24 up to Month 36 (DB treatment period for study 28981 (REFLEXION)
Population: DB Safety Population 28981 (REFLEXION) included all the participants who discontinued DB treatment in REFLEX study 27025 (NCT00404352) and were enrolled in 28981 (REFLEXION) study and received at least one dose of DB treatment in this study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (DB Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN]-beta-1a (RNF) injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first.
- RNF 44 Mcg Once Weekly (DB Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first.
- RNF 44 Mcg Thrice Weekly (DB Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 36 months or until conversion to CDMS whichever occurs first.
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) | RNF 44 Mcg Once Weekly (DB Population) | RNF 44 Mcg Thrice Weekly (DB Population)
Number analyzed (Participants) | 84 | 117 | 99
participants
  AEs | 79 | 67 | 45
  SAEs | 3 | 2 | 4
  AEs leading to discontinuation | 2 | 0 | 2

13. Secondary Outcome: Time to Conversion to Clinically Definite Multiple Sclerosis (CDMS) Defined by Either a Second Attack or a Sustained Increase (Greater Than or Equal to 1.5 Points) in the Expanded Disability Status Scale (EDSS) Score up to Month 60
Description: CDMS was defined by the occurrence of a second attack or relapse over 60 months in participants who presented with clinically isolated syndrome (CIS) accompanied by an abnormal magnetic resonance imaging (MRI) scan. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]) was calculated. Time to conversion to CDMS was represented by Kaplan-Meier estimates of the cumulative percentage (%) of participants with CDMS.
Time Frame: Baseline (Day 1 of Study 27025) up to 60 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cumulative % of participants with CDMS
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN]-beta-1a (RNF) injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first. After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months.
- RNF 44 Mcg Once Weekly (Integrated ITT Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months.
- RNF 44 Mcg Thrice Weekly (Integrated ITT Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months.
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
Cumulative % of participants with CDMS | 44.6 [36.6 to 52.6] | 40.7 [32.8 to 48.6] | 39.2 [30.8 to 47.6]

14. Secondary Outcome: Time to Confirmed Expanded Disability Status Scale (EDSS) Progression up to 60 Months
Description: as for outcome 2
Time Frame: Baseline (Day 1 of Study 27025) up to 60 Months
Population: as for outcome 1
Measure: Number; unit: % of participants with EDSS progression
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
% of participants with EDSS progression | 11.0 | 18.7 | 18.4

15. Secondary Outcome: Number of Combined Unique Active (CUA) Lesions, New Time Constant 2 (T2) Lesions, New Gadolinium Enhanced (Gd+) Lesions and New T1 Lesions Per Participant Per Scan at Month 60
Description: Number of CUA lesions, new T2 lesions, new Gd+ Lesions and new T1 lesions were measured by using MRI scans.
Time Frame: Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (ITT Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of RNF injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. 84 participants were initially assigned to DB RNF 44 mcg thrice weekly and 49 participants were initially assigned to OL RNF 44 mcg thrice weekly (4 participants from DB converted to CDMS and switched to OL period over course of this study)
- RNF 44 Mcg Once Weekly (ITT Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. 117 participants were initially assigned to DB RNF 44 mcg thrice weekly and 25 participants were initially assigned to OL RNF 44 mcg thrice weekly (10 participants from DB converted to CDMS and switched to OL period over course of this study)
- RNF 44 Mcg Thrice Weekly (ITT Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first. After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months. 99 participants were initially assigned to DB RNF 44 mcg thrice weekly and 28 participants were initially assigned to OL RNF 44 mcg thrice weekly (6 participants from DB converted to CDMS and switched to OL period over course of this study)
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (ITT Population) | RNF 44 Mcg Once Weekly (ITT Population) | RNF 44 Mcg Thrice Weekly (ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
lesions
  CUA Lesions (n=102, 121, 110) | 1.46 (3.394) | 1.60 (3.542) | 1.94 (4.803)
  New T2 Lesions (n=102, 121, 110) | 1.17 (2.576) | 1.17 (2.628) | 1.35 (3.284)
  New Gd+ Lesions (n=102, 121, 110) | 0.24 (0.823) | 0.36 (1.225) | 0.48 (1.618)
  New T1 Lesions (n=102, 120, 110) | 0.57 (1.656) | 0.69 (1.659) | 0.71 (1.917)

16. Secondary Outcome: Change From Baseline in Time Constant 1 (T1) Hypointense Volume, and Time Constant 2 (T2) Lesion Volume at Month 60
Description: Change from baseline in lesion volume was measured by using MRI scans for T1 hypointense lesions and T2 lesions.
Time Frame: Baseline (Day 1 of Study 27025), Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (ITT Population) | RNF 44 Mcg Once Weekly (ITT Population) | RNF 44 Mcg Thrice Weekly (ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
mm^3
  T1 lesion volume at Baseline (n=171,175,171) | 670.3 (1054.1) | 774.8 (1288.0) | 675.0 (1049.9)
  Change at Month 60 (n=102,120,110) | 415.0 (1080.3) | 412.3 (1020.8) | 261.8 (1006.1)
  T2 lesion volume at Baseline (n=171,175,171) | 3334.9 (3990.4) | 3853.1 (4716.7) | 3110.5 (3410.7)
  Change at Month 60 (n=102,121,110) | 119.4 (2225.2) | 25.0 (2827.1) | -188.5 (2576.1)

17. Secondary Outcome: Percent Change From Baseline in Brain Volume at Month 60
Description: Percent Change in brain volume was measured by using MRI scans.
Time Frame: Baseline (Day 1 of Study 27025), Month 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 98 | 120 | 110
percent change | -1.82 (1.494) | -1.54 (1.378) | -2.03 (1.644)

18. Secondary Outcome: Percentage of Participants With Conversion to McDonald Multiple Sclerosis (MS) at Month 60
Description: as for outcome 6
Time Frame: Month 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
percentage of participants | 84.2 | 82.9 | 72.5

19. Secondary Outcome: Change From Baseline in Paced Auditory Serial Addition Test 3 (PASAT-3) Score at Month 60
Description: The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Score ranges from '0-60'. Higher scores reflect better neurological function and a positive change from baseline indicates improvement.
Time Frame: Baseline (Day 1 of Study 27025), Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
units on a scale
  Baseline (n=171, 175, 171) | 0.0358 (0.8787) | -0.0909 (1.1223) | 0.0031 (1.1387)
  Change at Month 60 (n=112, 132, 118) | 0.4109 (0.6844) | 0.4785 (0.9886) | 0.4608 (0.8630)

20. Secondary Outcome: Percentage of Relapse-Free Participants at Month 60
Description: as for outcome 8
Time Frame: Month 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
percentage of participants | 34.5 | 45.1 | 40.9

21. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Month 60
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. The change in EDSS score at Month 60 was calculated as EDSS score at Month 60 minus EDSS score at baseline.
Time Frame: Baseline (Day 1 of Study 27025), Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
units on a scale
  Baseline (n=171,175,171) | 1.53 (0.77) | 1.50 (0.72) | 1.51 (0.83)
  Change at Month 60 (n=111,133,117) | -0.11 (0.94) | -0.01 (1.01) | 0.04 (1.02)

22. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score at Month 60
Description: as for outcome 10
Time Frame: Baseline (Day 1 of Study 27025), Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated ITT Population) | RNF 44 Mcg Once Weekly (Integrated ITT Population) | RNF 44 Mcg Thrice Weekly (Integrated ITT Population)
Number analyzed (Participants) | 171 | 175 | 171
Z-score
  MFSC score at Baseline (n=171,175,171) | 0.0352 (0.5844) | 0.0071 (0.6653) | -0.0575 (0.6226)
  Change at Month 60 (n=112,132,132) | 0.2290 (0.4824) | 0.2213 (0.5602) | 0.2192 (0.6229)

23. Secondary Outcome: Numbers of Participants With Binding Antibodies (BAb) and Neutralizing Antibody (NAb) at Month 60
Description: BAbs are all antibodies which are capable of binding to the RNF irrespective of their binding site. NAbs are defined as a subgroup of BAbs which bind to the active sites of the RNF and therefore neutralize its potency. NAbs were detected using a viral cytopathic assay. BAbs were measured by using an ELISA.
Time Frame: Month 60
Population: as for outcome 11
Measure: Number; unit: participants
Groups:
- Placebo/RNF 44 Mcg Thrice Weekly (Integrated DB Population): Participants who were initially randomized in study 27025 (REFLEX) to the placebo treatment group were switched to single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN]-beta-1a (RNF) injection administered subcutaneously 3 times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 60 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first.
- RNF 44 Mcg Once Weekly (Integrated DB Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first.
- RNF 44 Mcg Thrice Weekly (Integrated DB Population): Single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and then 44 mcg until 60 months or until conversion to CDMS whichever occurs first.
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (Integrated DB Population) | RNF 44 Mcg Once Weekly (Integrated DB Population) | RNF 44 Mcg Thrice Weekly (Integrated DB Population)
Number analyzed (Participants) | 115 | 130 | 115
participants
  BAb- | 89 | 99 | 100
  BAb+ | 25 | 30 | 15
  BAb (Missing) | 1 | 1 | 0
  NAb- | 97 | 110 | 102
  NAb+ | 18 | 20 | 13

24. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Treatment Discontinuation
Description: as for outcome 12
Time Frame: Month 24 up to Month 60
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) | RNF 44 Mcg Once Weekly (DB Population) | RNF 44 Mcg Thrice Weekly (DB Population)
Number analyzed (Participants) | 84 | 117 | 99
participants
  AEs | 70 | 96 | 84
  SAEs | 7 | 7 | 9
  AEs leading to discontinuation | 3 | 0 | 2

ADVERSE EVENTS:
Time Frame: Month 24 to 60 for both DB safety population and OL safety population
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) | RNF 44 Mcg Once Weekly (DB Population) | RNF 44 Mcg Thrice Weekly (DB Population) | Placebo/RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly | RNF 44 Mcg Once Weekly /OL RNF 44 Mcg Thrice Weekly | RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly
Serious Adverse Events (participants affected / at risk) | 7/84 | 7/117 | 9/99 | 2/58 | 3/51 | 4/46
Other Adverse Events (participants affected / at risk) | 69/84 | 97/117 | 84/99 | 46/58 | 37/51 | 36/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) (N=84) | RNF 44 Mcg Once Weekly (DB Population) (N=117) | RNF 44 Mcg Thrice Weekly (DB Population) (N=99) | Placebo/RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly (N=58) | RNF 44 Mcg Once Weekly /OL RNF 44 Mcg Thrice Weekly (N=51) | RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly (N=46)
Abscess intestinal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Endometritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Angina stable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Foetal chromosome abnormality (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/RNF 44 Mcg Thrice Weekly (DB Population) (N=84) | RNF 44 Mcg Once Weekly (DB Population) (N=117) | RNF 44 Mcg Thrice Weekly (DB Population) (N=99) | Placebo/RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly (N=58) | RNF 44 Mcg Once Weekly /OL RNF 44 Mcg Thrice Weekly (N=51) | RNF 44 Mcg Thrice Weekly/OL RNF 44 Mcg Thrice Weekly (N=46)
Leukopenia (Blood and lymphatic system disorders) | 9 | 2 | 2 | 0 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 4 | 1 | 5 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 3 | 5 | 0 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 1 | 5 | 2 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 8 | 3 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 5 | 4 | 4 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2
Influenza like illness (General disorders) | 45 | 39 | 17 | 11 | 12 | 10
Injection site erythema (General disorders) | 17 | 6 | 8 | 4 | 8 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 3 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 3
Bronchitis (Infections and infestations) | 3 | 5 | 6 | 4 | 1 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1
Influenza (Infections and infestations) | 3 | 8 | 7 | 4 | 2 | 3
Nasopharyngitis (Infections and infestations) | 12 | 14 | 9 | 6 | 7 | 4
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 10 | 11 | 10 | 6 | 5 | 5
Urinary tract infection (Infections and infestations) | 1 | 8 | 3 | 2 | 3 | 4
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 8 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 4 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 6 | 5 | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1 | 1
Headache (Nervous system disorders) | 11 | 19 | 16 | 4 | 6 | 9
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 3
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 7 | 4 | 2 | 0 | 3
Depression (Psychiatric disorders) | 1 | 6 | 2 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 1 | 7 | 4 | 2 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2 | 2
Hypertension (Vascular disorders) | 5 | 7 | 1 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to publish any results communication in connection with the study. The PI shall submit any communications including study results to the sponsor for review 30 working days prior to communication submission. The sponsor can request the PI to modify or delete any sponsor's proprietary information. If the PI refuses the modification, the submission shall be postponed for 60 days from PI refusal, to provide the sponsor the opportunity to file a patent or seek legal remedies.